CLINICAL TRIAL: NCT01719497
Title: Imaging of Cannabinoid 1 Receptors Using [11C]OMAR and PET
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 0906005296
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Obesity; Alcohol Dependence; High Stress
MeSH Terms: conditions — Obesity; Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Alcohol: Subjects diagnosed with alcohol dependence
  Interventions: Drug: [C-11]OMAR
- Obese: Subjects diagnosed with obesity
  Interventions: Drug: [C-11]OMAR
- High Stress: Subjects diagnosed with high stress
  Interventions: Drug: [C-11]OMAR
- Healthy: Subjects deemed medically healthy
  Interventions: Drug: [C-11]OMAR

INTERVENTIONS:
Drug: [C-11]OMAR — PET radioligand

SUMMARY:
The aim of the present study is to conduct a human trial of [C-11]OMAR, a new PET imaging agent for the brain cannabinoid type 1 receptors (CB1), to determine its pharmacokinetics and binding characteristics.

DETAILED DESCRIPTION:
This is a pilot, 2-part study to assess the kinetics of radioactivity in medically healthy subjects, subjects with alcohol dependency (AD), and obese subjects following the intravenous administration of the imaging agent [C-11]OMAR.

ELIGIBILITY:
Inclusion Criteria:

1. Are overtly healthy males or females (other than AD or obesity), as determined by medical history and physical examination. Males and females with stable medical problems that, in the investigator's opinion, will not significantly alter the disposition of the drug, will not place the subject at increased risk by participating in the study, and will not interfere with interpretation of the data.
2. Are between the ages of 18 and 65 years, inclusive.
3. Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator. (Note: specific laboratory tests are listed in section 3.4)
4. Have arterial access sufficient to allow blood sampling as per the protocol.
5. Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
6. Have given written informed consent approved by the ethical review board governing the site.

Exclusion Criteria:

1. Are currently enrolled in, or discontinued within the last [30 days] from, a clinical trial involving an off-label use of an investigational drug or device, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
2. Current substance abuse (other than AD) including marijuana use, or severe systemic disease based on history and physical exam.
3. Laboratory tests with clinically significant abnormalities or positive urine toxicology screen. (Note: specific laboratory tests are listed in section 3.4)
4. Prior participation in other research protocols in the last year such that radiation exposure would exceed the annual limits.
5. Presence of ferromagnetic metal in the body or heart pacemaker.
6. Are persons who have previously completed or withdrawn from this study or any other study investigating [C-11]OMAR.
7. Regularly use known drugs of abuse (other than alcohol) within 30 days of the study and/or show positive findings on urinary drug screening.
8. Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
9. Are women with a positive pregnancy test or women who are lactating.
10. Have a history of head trauma with prolonged loss of consciousness (>10 minutes), or any neurological condition including stroke or seizure (excluding a single childhood febrile seizure) or a history of migraine headaches
11. History of adverse drug reactions or intolerance to more than three types of systemically administered medications
12. Have used any prescription medication (except for oral contraceptives or hormone replacement therapy) or over-the-counter medication (including herbal remedies or diet aids) within 14 days of the imaging session. Multiple vitamins are specifically permitted
13. Have implanted or embedded metal objects or fragments in the head or body that would present a risk during the MRI scanning procedure, or have worked with ferrous metals either as a vocation or hobby (for example, as a sheet metal worker, welder, or machinist) in such a way that might have led to unknown, indwelling metal fragments that could cause injury if they moved in response to placement in the magnetic field
14. Have had exposure to ionizing radiation that in combination with the study tracer would result in a cumulative exposure that exceeds recommended exposure limits

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: N = 30 Medically Healthy control subjects N = 30 Subjects with high stress exposure N = 30 Subjects with Alcohol Dependence (AD) N = 30 Obese subjects
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2009-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
No outcome measures for this study, this is an imaging study only | Upon study completion

CONTACTS AND LOCATIONS:
Overall Officials: Marc N Potenza, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States